CLINICAL TRIAL: NCT00240734
Title: A Randomized, Double-blind, Placebo-Controlled Study Evaluating Weekly Epoetin Alfa (PROCRIT�) Administration on Hemoglobin Response and Safety in Diabetic Subjects With the Anemia of Chronic Kidney Disease (CKD)
Brief Title: Treatment of Anemia in Diabetic Subjects With CKD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was stopped for slow enrollment after enrolling only 11 of 180 patients in six months time.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004597
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Anemia
Keywords: Anemia; Chronic renal failure; pre-dialysis; diabetic
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to compare the proportion of subjects receiving either Epoetin alfa (PROCRITÂ®) or placebo who are able to achieve a hemoglobin response, defined by at least a 1 gram/deciliter increase from baseline by Week 17.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind, placebo controlled, multi-center study in diabetic subjects with the anemia of chronic kidney disease. Subjects will be randomly assigned in a 1:1 ratio to receive either Epoetin alfa (PROCRIT®) or matching placebo for sixteen weeks. Epoetin alfa (PROCRIT®) is indicated for the treatment of anemia associated with chronic renal failure (pre-dialysis), non-myeloid malignancies receiving chemotherapy, in HIV-infected subjects receiving zidovudine therapy, and in anemic subjects undergoing elective non-cardiac, non-vascular surgery to reduce the need for allogenic blood transfusion during high-volume blood loss procedures. This study is being undertaken to assess, under well-controlled conditions, the effect of weekly Epoetin alfa (PROCRIT®) treatment on hemoglobin response in diabetic subjects with the anemia of chronic kidney disease. The study hypothesis is that weekly PROCRIT treatment will be effective in achieving a hemoglobin response than placebo, where hemoglobin response is defined by at least a 1 gram/deciliter increase from baseline by Week 17. The subjects are administered study drug (PROCRIT® or matching placebo) once weekly by subcutaneous injection by a health care professional for 16 weeks. The initial dose of study drug is either PROCRIT® 10,000 U (1.0 mL) or matching placebo. The maximum dose administered is 20,000 U (2.0 mL).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of diabetes mellitus
* History of documented proteinuria or microalbuminuria
* A glomerular filtration rate between 15 and 90 mL/minute/1.73m2
* Subjects with hemoglobin greater than or equal to 9.0 /dL and less than or equal to 11.0 g/dL.

Exclusion Criteria:

* A current diagnosis of poorly controlled high blood pressure (hypertension) (systolic blood pressure > 150 mm Hg or diastolic blood pressure > 100 mm Hg) after adequate anti hypertensive therapy
* Subjects with severe neuropathy or peripheral vascular disease with gait instability
* Subjects scheduled to receive dialysis during the course of the study
* Subjects with a transferrin saturation < 20% or ferritin level < 50 ng/dL
* Subjects with active malignancy, defined as a malignancy requiring current therapy (surgery, chemotherapy, or radiotherapy) or a history of treatment for malignancy in the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-03; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the hemoglobin response rate, defined as the proportion of subjects who achieve at least a 1 gram per deciliter hemoglobin increase from baseline by Week 17.

SECONDARY OUTCOMES:
The secondary endpoints include evaluation of health-related quality life, hemoglobin change over time, time to hemoglobin response, and transfusion utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- See also: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating Weekly PROCRIT (Epoetin alfa) Administration on Hemoglobin Response and Safety in Diabetic Subjects with the Anemia of Chronic Kidney Disease (CKD) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=603&filename=CR004597_CSR.pdf